CLINICAL TRIAL: NCT05317195
Title: A Single-center, Randomized, Controlled, Open-label Study to Investigate the Nicotine Pharmacokinetic Profiles and Subjective Effects of Four Variants of Nicotine Pouch 1.0 Compared to Velo® Ice Cool and Zyn® Cool Mint Mini Dry in Healthy Smokers
Brief Title: Nicotine Pharmacokinetics and Subjective Effects of Nicotine Pouch 1.0 Compared to Velo® Ice Cool and Zyn® Cool Mint Mini Dry in Healthy Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P5-PK-01-EXP
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Smoking; Nicotine
Keywords: Nicotine-containing products; Nicotine delivery
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- NP-1 (Experimental): Nicotine Pouch 1.0 (variant NP-1)
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP
- NP-2 (Experimental): Nicotine Pouch 1.0 (variant NP-2)
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP
- NP-3 (Experimental): Nicotine Pouch 1.0 (variant NP-3)
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP
- NP-4 (Experimental): Nicotine Pouch 1.0 (variant NP-4)
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP
- Velo-NP (Active Comparator): Velo® Ice Cool
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP
- Zyn-NP (Active Comparator): Zyn® Cool Mint Mini Dry
  Interventions: Other: NP-1; Other: NP-2; Other: NP-3; Other: NP-4; Other: Velo-NP; Other: Zyn-NP

INTERVENTIONS:
Other: NP-1 — NP-1; 8.4 mg nicotine; pH 8.0; moisture 30
Other: NP-2 — NP-2; 8.4 mg nicotine; pH 9.0; moisture 30
Other: NP-3 — NP-3; 3.6 mg nicotine; pH 8.0; moisture 15
Other: NP-4 — NP-4; 3.6 mg nicotine; pH 8.0; moisture 30
Other: Velo-NP — Velo-NP; 10 mg nicotine;
Other: Zyn-NP — Zyn-NP; 3 mg nicotine;

SUMMARY:
This is a single-center, randomized, controlled, open-label, cross-over study in healthy smoking subjects to investigate the nicotine pharmacokinetic (PK) profiles of 4 variants of Nicotine pouch 1.0 compared to marketed Velo - Nicotine Pouch (NP) and Zyn-NP. In addition, pharmacodynamic (PD) effects will be evaluated to provide further insights on Nicotine pouch 1.0 product acceptance and abuse liability. The study will be conducted with 3 periods and 6 sequences in a Williams design (cross-over).

DETAILED DESCRIPTION:
Study Title:

Nicotine Pharmacokinetics and Subjective Effects of Nicotine Pouch 1.0 Compared to Velo® Ice Cool and Zyn® Cool Mint Mini Dry in Healthy Smokers

Who carried out the research? This research was sponsored and funded by Philip Morris Products S.A.

What public involvement there was in the study? The study recruited 31 healthy adults who were currently smoking.

Where and when the study took place The study was conducted at a clinical trial facility managed by a contract research organization in Belfast, Northern Ireland, from March 15th to August 18th 2022.

Why was the research needed? The research was needed to understand the pharmacokinetic profiles of four variants of a nicotine pouch.

What were the main questions studied? The study measured the nicotine absorption of the four variants of nicotine pouch (NP-1; NP-2; NP-3; NP-4) together with two nicotine pouches marketed by other companies (Zyn-NP and Velo-NP). Participants were also asked to evaluate their experience of using the nicotine pouches.

Who participated in the study? The study recruited 31 healthy, male or female, adults aged between 21 and 65 years who were currently smoking. The subjects did not plan to quit using tobacco and/or nicotine products within the next 3 months and had smoked continuously for at least the last 3 years prior to joining the study..

Each subject was given full and adequate oral and written information about the nature, purpose, possible risks and benefits of the study. Once each subject had received all the necessary information, and if he/she agreed to participate, this was documented in an Informed Consent Form with the date, time and signature of both the subject and the Investigator.

Subjects were informed that they were free to withdraw from the study at any time.

What treatments or interventions did the participants take/receive? The participants were requested to use a tobacco-free nicotine pouch for a period of 30 minutes. Blood samples were taken before, during, and after the product use period.

Participants were also asked to evaluate their experience of using the nicotine pouches, using the Product Evaluation Scale (PES).

The PES is composed of seven items which address the degree to which subjects experience seven different effects (Product Satisfaction, Psychological Rewards, Aversion, Craving Relief, Easy to Use, Comfortable Using, Concerned about Dependence) as a result of using the investigational products, rated on a 7 point scale from 1 = "not at all" to 7 = "extremely."

What happened during the study? The study was conducted with six periods and six sequences in a cross-over design. On Day -1, subjects were randomized to one of the six study sequences.

After enrollment, subjects performed a product test with Nicotine Pouch 1.0 (NP-1) for 30 minutes (± 1 minute). One NP-1 nicotine pouch was placed between the upper lip and the gum for 30 minutes and subjects were instructed not to manipulate the pouch with the tongue or lips.

After the product test, subjects were required to abstain from any nicotine/tobacco-containing product use until the first product use on Day 1.

On Day 1 to Day 3, after at least 8 hours of abstinence from any nicotine/tobacco-containing products (nicotine wash-out), subjects used one variant of NP 1.0, Velo-NP, or Zyn-NP according to the randomized product use sequence for 30 minutes (± 1 minute). The used NP were collected for long-term storage to determine the residual nicotine after product use to estimate the amount of nicotine delivered during the 30-minute use period.

Subjects completed questionnaires about product evaluation, craving, and liking assessments.

In the morning on Day 1, 12 blood samples were collected for determination of nicotine concentration. Additional blood samples were taken for determination of the nicotine concentration on Day 2 and Day 3.

After Discharge at Day 3, the subjects entered a 3-day Safety Follow-Up period during which adverse reactions associated with product use reported by the subjects were collected and the follow-up of any ongoing adverse reactions was conducted by the study investigational site.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject has smoked continuously for at least the last 3 years prior to the Screening visit.
* Subject has smoked ≥ 10 commercially available cigarettes per day for 4 weeks prior to Screening Visit and Admission. Smoking status will be verified based on a urinary cotinine test (cotinine ≥ 500 ng/mL).
* Subject does not plan to quit using tobacco and/or nicotine products within the next 3 months.
* Smoking, healthy subject as judged by the Investigator or designee based on available assessments from the Screening period.

Main Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason other than medical.
* Subject is legally incompetent, or physically or mentally incapable of giving consent.
* Subject has a clinically relevant disease that requires medication, which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject has donated or received whole blood or blood products within 30 days prior to Screening Visit.
* Subject has a BMI < 18.5 kg/m2 or > 32.0 kg/m2 (Europe) or > 35.0 kg/m2 (USA).
* For women only: subject is pregnant (does not have negative pregnancy test at Screening Visit and at Admission) or is breastfeeding.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajkumar Chetty, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 subjects were enrolled in the study, which was conducted at a clinical trial facility managed by a contract research organization.
Pre-assignment Details: Of the 31 enrolled subjects who performed a product test, 24 were randomized to product use. Seven of the 31 enrolled subjects were not randomized because only 24 subjects were required for the study.
Groups:
- All Study Participants: All study participants.
Period: Product Test (Enrolled Subjects)
Arm/Group | All Study Participants
Started | 31
Completed | 31
Not Completed | 0
Period: Randomization
Arm/Group | All Study Participants
Started | 31
Completed | 24
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Discontinued | 6
Period: Admission
Arm/Group | All Study Participants
Started | 24
Completed | 22
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Product Use (Randomized Subjects)
Arm/Group | All Study Participants
Started | 22
NP-1 | 22
NP-2 | 22
NP-3 | 22
NP-4 | 22
Velo-NP | 22
Zyn-NP | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: The safety population was a subset of the screened population and comprised all the subjects who signed ICF consent and had at least one exposure to NP 1.0 (including the product test with NP-1 at Admission).
Arm/Group | Safety Population
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Fagerström score [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a standard instrument for assessing nicotine dependence. Subjects respond to six items in a questionnaire to obtain a total score between 0 and 10. Higher scores indicate an increased level of nicotine dependence.
  units on a scale | 5.2 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Background-corrected Maximum Plasma Concentration [Cmax]
Description: To measure the background-corrected maximum plasma concentration [Cmax] of 4 variants of NP 1.0 nicotine pouches compared to Velo-NP and Zyn-NP in healthy smokers from a 30 minutes product use period.
Time Frame: T0 = start of product use. Blood was drawn 5 minutes prior to T0, and then 5, 10, 15, 20, 25, 30, 35, 40 minutes, 1, 3, and 6 hours after T0, on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon).
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 21 | 22 | 22 | 22 | 22
ng/mL | 8.109 [6.570 to 9.649] | 11.48 [9.544 to 13.42] | 2.629 [1.670 to 3.588] | 3.464 [2.929 to 3.999] | 11.32 [9.880 to 12.75] | 9.257 [8.066 to 10.45]

2. Primary Outcome: Background-corrected Time to the Maximum Concentration [Tmax]
Description: To measure the background-corrected time to the maximum concentration [Tmax] of 4 variants of NP 1.0 nicotine pouches compared to Velo-NP and Zyn-NP in healthy smokers from a 30 minutes product use period.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 21 | 22 | 22 | 22 | 22
minutes | 35.70 [10.1 to 179] | 34.80 [9.96 to 60.4] | 34.89 [9.72 to 60.7] | 34.98 [29.8 to 64.3] | 33.99 [9.72 to 180] | 34.95 [22.9 to 59.7]

3. Primary Outcome: Area Under the Background-corrected Concentration-time Curve (AUC) From Start of Product Use, Extrapolated to Infinity (AUC Infinity)
Description: To measure the area under the background-corrected concentration-time curve (AUC) from start of product use of 4 variants of NP 1.0 nicotine pouches compared to Velo-NP and Zyn-NP in healthy smokers from a 30 minutes product use period.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: min*ng/mL
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 21 | 22 | 22 | 22 | 22
min*ng/mL | 128.2 [97.73 to 158.6] | 217.3 [177.6 to 256.9] | 41.35 [28.28 to 54.42] | 49.30 [40.87 to 57.73] | 201.3 [173.9 to 228.7] | 136.0 [112.6 to 159.3]

4. Secondary Outcome: Score of Cigarette Craving by the Visual Analog Scale (VAS)-Craving Assessment
Description: To measure cigarette craving by the visual analog scale (VAS)-craving assessment in healthy smokers following a 30 minutes product use period of 4 variants of Nicotine pouch 1.0 compared to Velo-NP and Zyn-NP. Craving was assessed at selected time points on a scale from "no craving" (0 mm) to "strong craving" (100 mm) by measuring the number of millimeters (0-100 mm) from the "no craving" point to the point at which the drawn line intersected the scale.
Time Frame: Measured before, and up to 6 hours post-product use on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
score on a scale
  Pre-Product Use | 61.0 [46.7 to 75.2] | 62.6 [49.6 to 75.6] | 64.3 [51.4 to 77.1] | 67.4 [55.0 to 79.8] | 68.6 [56.8 to 80.4] | 68.9 [54.9 to 82.8]
  5 min Post-Product Use | 38.5 [26.5 to 50.6] | 38.1 [26.5 to 49.7] | 50.3 [38.2 to 62.5] | 42.6 [30.8 to 54.4] | 38.7 [26.8 to 50.7] | 39.4 [25.7 to 53.1]
  10 min Post-Product Use | 36.4 [23.1 to 49.7] | 33.8 [22.1 to 45.5] | 43.0 [29.9 to 56.1] | 38.6 [26.9 to 50.3] | 34.3 [23.2 to 45.5] | 29.0 [18.1 to 40.0]
  15 min Post-Product Use | 27.3 [16.8 to 37.7] | 29.9 [17.7 to 42.1] | 39.5 [26.4 to 52.6] | 36.5 [23.8 to 49.3] | 31.7 [21.1 to 42.3] | 26.9 [15.8 to 37.9]
  20 min Post-Product Use | 29.2 [18.5 to 39.9] | 31.7 [19.2 to 44.3] | 38.0 [24.8 to 51.2] | 36.4 [23.8 to 48.9] | 26.9 [16.4 to 37.3] | 22.7 [12.6 to 32.8]
  25 min Post-Product Use | 29.1 [18.2 to 40.1] | 28.6 [17.3 to 39.8] | 46.1 [32.3 to 59.9] | 35.8 [24.4 to 47.3] | 24.1 [14.6 to 33.5] | 20.0 [11.8 to 28.3]
  30 min Post-Product Use | 28.8 [17.0 to 40.6] | 28.3 [17.1 to 39.5] | 37.2 [24.3 to 50.0] | 35.4 [23.5 to 47.3] | 24.2 [13.7 to 34.8] | 19.5 [10.4 to 28.7]
  35 min Post-Product Use | 27.2 [16.2 to 38.1] | 27.1 [16.0 to 38.2] | 36.9 [23.5 to 50.2] | 33.7 [21.0 to 46.4] | 23.4 [13.5 to 33.2] | 19.5 [9.7 to 29.3]
  40 min Post-Product Use | 29.0 [17.2 to 40.9] | 29.5 [18.3 to 40.7] | 34.6 [22.2 to 46.9] | 33.5 [20.5 to 46.5] | 22.8 [13.0 to 32.6] | 21.1 [11.4 to 30.9]
  1 hr Post-Product Use | 26.8 [15.8 to 37.7] | 32.0 [20.3 to 43.7] | 44.9 [31.4 to 58.4] | 35.8 [23.6 to 48.0] | 24.3 [14.4 to 34.3] | 24.7 [14.5 to 34.9]
  3 hr Post-Product Use | 45.8 [31.3 to 60.3] | 52.8 [40.4 to 65.3] | 53.9 [41.5 to 66.2] | 51.5 [38.3 to 64.7] | 42.1 [30.1 to 54.2] | 48.4 [34.7 to 62.0]
  6 hr Post-Product Use | 58.3 [44.5 to 72.1] | 60.1 [46.1 to 74.1] | 64.2 [50.4 to 77.9] | 57.8 [45.0 to 70.6] | 57.0 [43.0 to 70.9] | 54.2 [39.9 to 68.5]

5. Secondary Outcome: Score of "in the Moment" Product Liking by the VAS-liking Assessment
Description: To measure "in the moment" product liking by the VAS-liking assessment in healthy smokers following a 30 minutes product use period of 4 variants of Nicotine pouch 1.0 compared to Velo-NP and Zyn-NP. Product liking was assessed at selected time points on a scale from "strong disliking" (0 mm) to "strong liking" (100 mm) by measuring the number of millimeters (0-100 mm) from the "strong disliking" point to the point at which the drawn line intersected the scale.
Time Frame: Measured up to 1 hour post-product use on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
score on a scale
  5 min Post-Product Use | 49.7 [39.6 to 59.8] | 55.8 [48.2 to 63.5] | 50.1 [41.0 to 59.2] | 48.2 [39.3 to 57.1] | 51.7 [44.3 to 59.1] | 60.2 [51.9 to 68.5]
  10 min Post-Product Use | 54.8 [43.7 to 65.8] | 56.2 [45.7 to 66.7] | 52.1 [42.8 to 61.4] | 52.1 [42.8 to 61.5] | 55.8 [47.1 to 64.5] | 60.6 [50.0 to 71.2]
  15 min Post-Product Use | 59.2 [49.0 to 69.5] | 57.2 [45.5 to 68.9] | 52.4 [41.7 to 63.1] | 52.7 [43.9 to 61.5] | 56.1 [46.7 to 65.5] | 58.7 [47.2 to 70.3]
  20 min Post-Product Use | 51.5 [39.7 to 63.2] | 53.8 [41.6 to 66.0] | 52.1 [41.4 to 62.8] | 54.5 [45.4 to 63.7] | 58.7 [47.1 to 70.3] | 60.3 [47.7 to 72.9]
  25 min Post-Product Use | 54.6 [42.5 to 66.8] | 54.0 [42.4 to 65.7] | 51.4 [39.7 to 63.1] | 52.7 [43.3 to 62.2] | 54.7 [41.0 to 68.4] | 61.6 [49.7 to 73.5]
  30 min Post-Product Use | 60.0 [48.1 to 71.8] | 53.5 [40.5 to 66.5] | 52.0 [41.5 to 62.6] | 51.7 [41.1 to 62.3] | 57.7 [44.8 to 70.7] | 59.9 [47.5 to 72.3]
  35 min Post-Product Use | 55.2 [42.6 to 67.8] | 56.5 [44.9 to 68.1] | 51.4 [40.4 to 62.3] | 54.0 [43.8 to 64.2] | 57.0 [44.4 to 69.6] | 59.4 [45.6 to 73.2]
  40 min Post-Product Use | 56.7 [44.0 to 69.4] | 54.2 [42.0 to 66.4] | 51.4 [40.3 to 62.6] | 53.6 [43.0 to 64.3] | 57.2 [45.2 to 69.3] | 58.7 [45.7 to 71.7]
  1 hr Post-Product Use | 54.7 [41.8 to 67.6] | 54.5 [43.0 to 65.9] | 49.8 [39.1 to 60.4] | 53.4 [43.5 to 63.2] | 55.6 [43.7 to 67.6] | 58.2 [45.9 to 70.5]

6. Secondary Outcome: Score of Overall Product Liking by the VAS-liking Assessment
Description: To measure overall product liking by the VAS-liking assessment in healthy smokers following a 30 minutes product use period of 4 variants of Nicotine pouch 1.0 compared to Velo-NP and Zyn-NP. Overall product liking was assessed at selected time points on a scale from "strong disliking" (0 mm) to "strong liking" (100 mm) by measuring the number of millimeters (0-100 mm) from the "strong disliking" point to the point at which the drawn line intersected the scale.
Time Frame: Measured after 30 minutes product use on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
score on a scale | 56.5 [46.8 to 66.3] | 53.2 [44.6 to 61.8] | 49.0 [40.1 to 57.9] | 49.5 [40.2 to 58.9] | 49.9 [39.3 to 60.5] | 52.3 [40.7 to 64.0]

7. Secondary Outcome: Score of Product Satisfaction by the VAS-satisfaction Assessment
Description: To measure product satisfaction by the VAS-satisfaction assessment in healthy smokers following a 30 minutes product use period of 4 variants of Nicotine pouch 1.0 compared to Velo-NP and Zyn-NP. Product satisfaction was was assessed at selected time points on a scale from "not at all" (0 mm) to "extremely" (100 mm) by measuring the number of millimeters (0-100 mm) from the "not at all" point to the point at which the drawn line intersected the scale.
Time Frame: Measured on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
score on a scale
  5 min Post-Product Use | 52.5 [42.3 to 62.6] | 51.5 [41.0 to 62.0] | 45.8 [35.8 to 55.8] | 50.2 [41.2 to 59.2] | 48.4 [39.9 to 56.9] | 55.8 [45.2 to 66.3]
  10 min Post-Product Use | 58.0 [46.6 to 69.3] | 57.4 [46.5 to 68.4] | 48.2 [37.4 to 59.1] | 50.0 [39.9 to 60.2] | 54.5 [45.1 to 63.8] | 62.0 [52.0 to 72.1]
  15 min Post-Product Use | 60.9 [50.9 to 70.8] | 57.9 [46.3 to 69.5] | 50.5 [40.3 to 60.8] | 49.5 [39.4 to 59.5] | 57.5 [48.4 to 66.7] | 62.4 [50.1 to 74.7]
  20 min Post-Product Use | 61.1 [50.4 to 71.9] | 52.0 [38.3 to 65.8] | 49.7 [39.0 to 60.4] | 49.3 [38.5 to 60.1] | 61.0 [49.4 to 72.6] | 65.2 [53.3 to 77.1]
  25 min Post-Product Use | 54.2 [41.3 to 67.1] | 56.8 [46.0 to 67.7] | 50.1 [38.8 to 61.4] | 50.8 [39.8 to 61.7] | 58.2 [45.7 to 70.6] | 67.5 [55.7 to 79.2]
  30 min Post-Product Use | 60.6 [47.5 to 73.6] | 58.2 [46.8 to 69.7] | 50.4 [39.4 to 61.4] | 50.2 [38.4 to 62.0] | 61.6 [49.2 to 74.0] | 67.3 [54.8 to 79.8]
  35 min Post-Product Use | 61.2 [49.9 to 72.5] | 56.0 [44.2 to 67.9] | 46.0 [34.6 to 57.5] | 52.9 [41.4 to 64.4] | 60.4 [48.4 to 72.4] | 65.1 [53.4 to 76.9]
  40 min Post-Product Use | 59.0 [45.9 to 72.2] | 53.2 [40.1 to 66.3] | 44.4 [31.8 to 57.0] | 51.7 [39.4 to 63.9] | 61.4 [51.0 to 71.8] | 60.5 [47.8 to 73.1]
  1 hr Post-Product Use | 54.2 [40.5 to 67.8] | 52.6 [40.3 to 65.0] | 43.5 [31.5 to 55.6] | 50.3 [38.9 to 61.8] | 57.9 [46.4 to 69.4] | 59.5 [47.4 to 71.5]
  3 hr Post-Product Use | 46.2 [34.5 to 58.0] | 37.3 [27.2 to 47.4] | 36.9 [26.3 to 47.5] | 37.3 [27.1 to 47.6] | 44.4 [33.2 to 55.5] | 38.1 [25.0 to 51.3]
  6 hr Post-Product Use | 32.6 [21.0 to 44.2] | 26.7 [15.4 to 38.0] | 33.6 [23.0 to 44.2] | 33.2 [23.3 to 43.1] | 29.2 [19.7 to 38.7] | 35.4 [23.0 to 47.7]

8. Secondary Outcome: Score of Product Intention to Use Again by the VAS-intention to Use Again Assessment
Description: To measure intention to use product again by the VAS-intention to use again assessment in healthy smokers following a 30 minutes product use period of 4 variants of Nicotine pouch 1.0 compared to Velo-NP and Zyn-NP. Intention to use again was was assessed at selected time points on a scale from "very unlikely" (0 mm) to "very likely" (100 mm) by measuring the number of millimeters (0-100 mm) from the "very unlikely" point to the point at which the drawn line intersected the scale.
Time Frame: Measured on day 1 (morning/afternoon), day 2 (morning/afternoon), and day 3 (morning/afternoon)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NP-1 | NP-2 | NP-3 | NP-4 | Velo-NP | Zyn-NP
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
score on a scale
  30 min Post-Product Use | 51.3 [37.7 to 64.9] | 52.0 [38.8 to 65.1] | 46.7 [35.1 to 58.2] | 48.3 [36.2 to 60.3] | 55.3 [42.9 to 67.6] | 57.9 [43.2 to 72.6]
  3 hr Post-Product Use | 48.8 [35.6 to 61.9] | 48.1 [37.8 to 58.4] | 51.6 [42.5 to 60.6] | 44.5 [33.0 to 55.9] | 50.9 [39.5 to 62.2] | 49.5 [35.3 to 63.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 27 days.
Description: Note that the "Safety Population (NP-1)" comprised 31 subjects who were enrolled in the study and performed a product test with NP-1 at admission. Following the product test, 24 subjects were randomized to product use.
Groups:
- Safety Population (NP-1 Test): Comprised all enrolled subjects who, on Day -1, performed a product test using NP-1 for 30 minutes (± 1 minute).
- Safety Population (NP-1): Comprised all enrolled subjects who were exposed to NP-1 during the study.
- Safety Population (NP-2): Comprised all enrolled subjects who were exposed to NP-2 during the study.
- Safety Population (NP-3): Comprised all enrolled subjects who were exposed to NP-3 during the study.
- Safety Population (NP-4): Comprised all enrolled subjects who were exposed to NP-4 during the study.
- Safety Population (Velo-NP): Comprised all enrolled subjects who were exposed to Velo-NP during the study.
- Safety Population (Zyn-NP): Comprised all enrolled subjects who were exposed to Zyn-NP during the study.
Arm/Group | Safety Population (NP-1 Test) | Safety Population (NP-1) | Safety Population (NP-2) | Safety Population (NP-3) | Safety Population (NP-4) | Safety Population (Velo-NP) | Safety Population (Zyn-NP)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/31 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05317195/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05317195/SAP_001.pdf